CLINICAL TRIAL: NCT03945643
Title: Is Blood Flow Through IPAVA and PFO Related to Breath-hold and SCUBA Diving-induced Pulmonary Hypertension?
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 07302018.031
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Patent Foramen Ovale; Intrapulmonary Arteriovenous Anastamosis
MeSH Terms: conditions — Foramen Ovale, Patent | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Breath hold divers will be administered sildenafil and placebo. Age-matched controls will be administered sildenafil and placebo.
Who Masked: Participant, Outcomes Assessor
Masking Description: Utilization of placebo to mask drug administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil administration (Active Comparator): Administration of 50mg sildenafil one time, one hour prior to measurements
  Interventions: Drug: Sildenafil
- Placebo administration (Placebo Comparator): Administration of 50mg placebo one time, one hour prior to measurements
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil — 50mg administration of sildenafil, one time, one hour prior to measurements.
  Arms: Sildenafil administration
Other: Placebo — 50mg administration in gel-encapsulated microcrystalline cellulose one time, one hour prior to measurements.
  Arms: Placebo administration

SUMMARY:
In summary, the investigators propose to study elite Croatian breath-hold and SCUBA divers. The investigators will quantify breath-hold hypoxia- and SCUBA diving-induced pulmonary hypertension and right heart function to investigate the relationships between PFO and IPAVA blood flow. The investigators will use a placebo-controlled intervention (sildenafil) to reduce pulmonary arterial pressure in these subjects to examine the impact of the change in pressure (or absence of change) on the relationships determined above.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (increased lung blood pressure) is a multifactorial disease without a cure. Investigating reversible forms of pulmonary hypertension induced under extreme conditions such as a prolonged breath-hold and/or SCUBA diving may help to better understand why some individuals develop this devastating disease, and others do not.

Pulmonary arterial pressure is typically very low in healthy humans. Low oxygen levels (hypoxia) cause a constriction of the lung blood vessels resulting in smaller diameters, but lung blood flow stays constant or increases. Having constant flow with smaller vessel diameters causes pulmonary arterial pressure to increase but it will return to normal once normal oxygen levels are restored. Moreover, there is an association with patent foramen ovale (PFO, small hole between the atria in the heart) and excessive pulmonary arterial pressures in low oxygen conditions. However, the reasons for the exacerbated increase in pulmonary arterial pressure in these subjects with a PFO (PFO+) is unknown, but may be due to an exaggerated constriction response to low oxygen.

During a breath-hold, the oxygen in the lung decreases and in elite breath-hold divers, it decreases to very low levels. Compared to subjects without a PFO (PFO-), the oxygen may drop even lower in those PFO+ subjects because deoxygenated blood travels through the small hole to mix with oxygenated blood, exacerbating the level to which blood oxygen decreases. Thus, using a breath-hold model of lung hypoxia is one approach to examining a hypoxia-induced increase in pulmonary arterial pressure - a method critically dependent upon the elite breath-hold diver's ability to hold their breath for significant durations.

Intrapulmonary arteriovenous anastomoses (IPAVA) are vessels within the lung that bypass capillaries. The investigator's group has investigated the possible roles these unique vessels may have in physiological and pathophysiological conditions. The investigators have found that IPAVA blood flow occurs when healthy subjects breathe low oxygen gas. The investigators have also found that IPAVA blood flow is inversely related to pulmonary arterial pressure. Specifically, individuals with high pulmonary arterial pressures have low IPAVA blood flow and vice versa.

The right ventricle of the heart pumps blood through the pulmonary artery to the lungs. Under resting conditions the right heart performs a minimal amount of work because the pressure in the lung blood vessels is low. When pulmonary arterial pressure increases, the work of the right side of the heart has to increase substantially to keep blood pumping through the lung. Thus, high pulmonary arterial pressures will increase the work of the right heart and may lead to right heart dysfunction thereby limiting the amount of blood the heart can pump. If the pressure is high enough to limit the amount of blood flowing through the lung then this can be detected by a reduction in pulmonary blood flow and/or changes in the function of the heart during contraction (systole) and relaxation (diastole). Accordingly, an intervention that reduces pulmonary arterial pressures during a breath-hold may have a beneficial effect on right heart function.

Taken together, during an elite breath-hold dive, where the level of oxygen decreases, the investigators expect that pulmonary arterial pressures will increase as lung oxygen levels decrease, and the reduction in oxygen may be even lower in PFO+ subjects. Furthermore, as blood oxygen levels decrease, IPAVA blood flow will increase in some PFO- subjects thereby keeping pulmonary arterial pressures low in those individuals. Conversely, PFO+ subjects and those PFO- subjects with low levels of IPAVA blood flow would be expected to have the greatest pulmonary pressures. Whether or not this is true is unknown. Therefore, Objective #1 will quantify pulmonary arterial pressure and right heart function and investigate their relationships with PFO and IPAVA blood flow in elite breath-hold divers while breathing concentrations of oxygen and carbon dioxide that mimic breath-hold-induced hypoxia [NOTE: it is not possible to image the heart during a breath hold because the fully inflated lung obstructs the ultrasound view of the heart]. Objective #2 will use sildenafil, a drug that increases nitric oxide bioavailability to dilate lung blood vessels, to decrease pulmonary arterial pressure while breathing concentrations of oxygen and carbon dioxide that mimic breath-hold-induced hypoxia. Investigators will quantify the effect of sildenafil on pulmonary arterial pressure and right heart function and will determine if it alters the relationship with IPAVA and PFO blood flow. As mentioned above, because those PFO+ subjects may have an exaggerated pulmonary vasoconstrictor response to hypoxia, sildenafil may be either less effective or ineffective in reducing the pulmonary arterial pressure in these subjects. Objective #3 will compare the elite breath hold diver study data to data obtained in age, sex and PFO matched subjects who do not have extensive experience with breath hold diving. To do this control subjects will undergo the same procedures in Objectives #1 & 2 above. These studies will also allow investigators to determine if there are differences in pulmonary vascular responses to hypoxia between those with and without breath hold diving experience.

In addition to the heart and lung alterations that occur in breath hold divers outlined above, it is also known that pulmonary arterial pressure increases after SCUBA diving, but returns to normal within a few hours. The mechanisms responsible for the increase in pulmonary arterial pressure are unknown, but are independent of hypoxia. Thus, investigating the relationship between IPAVA, PFO and SCUBA diving-induced increases in pulmonary arterial pressures offers an additional avenue for understanding pulmonary arterial hypertension susceptibility. Although it is unknown why pulmonary arterial pressure increases with SCUBA diving, it is known that pulmonary hypertension may contribute to right heart dysfunction and pulmonary edema (lung water accumulation) that can occur in subjects who are swimming and/or SCUBA diving. Prevention of increased pulmonary arterial pressures during and/or after a dive may help to prevent excessive right heart dysfunction and pulmonary edema. Thus, Objective #4 will quantify pulmonary arterial pressure and right heart function and investigate their relationships with PFO and IPAVA blood flow, pre- and post-SCUBA diving. Objective #5 will quantify the effect of sildenafil (post dive) on pulmonary arterial pressure and right heart function and will determine if it alters the relationship with IPAVA and PFO blood flow, pre- and post-SCUBA diving.

In summary, the investigators propose to study elite Croatian breath-hold and SCUBA divers. Investigators will quantify breath-hold hypoxia- and SCUBA diving-induced pulmonary hypertension and right heart function to investigate the relationships between PFO and IPAVA blood flow. Investigators will use a placebo-controlled intervention (sildenafil) to reduce pulmonary arterial pressure in these subjects to examine the impact of the change in pressure (or absence of change) on the relationships determined above.

ELIGIBILITY:
Inclusion Criteria:

* Reside in geographic location near Split, Croatia
* Elite breath hold divers
* Experienced SCUBA divers

Exclusion Criteria:

* Previous history of coronary artery disease
* Currently taking medication or herbal supplement for any heart or respiratory disease that cannot be ceased for 48 hours prior to testing
* Women who are pregnant or trying to become pregnant
* Previous history of any condition that would prevent the subject from performing a breath hold
* Taking sildenafil or products similar to sildenafil
* Taking Nitrates or other nitric oxide donors
* Control breath hold divers can't have previous breath hold diving experience

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary Pressure | 1 hour post intervention
  Pulmonary arterial pressure measured by ultrasound techniques
Concentration of Myoglobin | 1 hour post intervention
  Inflammatory cytokine
Concentration of MRP8/14 | 1 hour post intervention
  Inflammatory cytokine
Concentration of NGAL | 1 hour post intervention
  Inflammatory cytokine
Concentration Of CRP | 1 hour post intervention
  Inflammatory cytokine
Concentration Of MMP-2 | 1 hour post intervention
  Inflammatory cytokine
Concentration of OPN | 1 hour post intervention
  Inflammatory cytokine
Concentration Of SAA | 1 hour post intervention
  Inflammatory cytokine
Concentration of IGFBP-4 | 1 hour post intervention
  Inflammatory cytokine
Concentration of ICAM-1 | 1 hour post intervention
  Inflammatory cytokine
Concentration of VCAM-1 | 1 hour post intervention
  Inflammatory cytokine
Concentration of MMP-9 | 1 hour post intervention
  Inflammatory cytokine
Concentration of Cystatin C | 1 hour post intervention
  Inflammatory cytokine
Change in Q-IPAVA | 1 hour post intervention
  Minute bloodflow through intrapulmonary arteriovenous anastamoses

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lovering, PhD, Principal Investigator — University of Oregon
Locations (1):
- Cardiorespiratory and Pulmonary Physiology Lab, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Plan to not share IPD.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT03945643/Prot_SAP_002.pdf
  • Informed Consent Form (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT03945643/ICF_003.pdf